CLINICAL TRIAL: NCT05400278
Title: Characterizing the Genotype, Phenotype, Health Issues, and Quality of Life in Adults With Bardet-Biedl Syndrome
Brief Title: Characterizing the Genotype and Phenotype in Adults With Bardet-Biedl Syndrome
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Lovisenberg Diakonale Hospital (Other); Sykehuset Telemark (Other Government)
Responsible Party: Principal Investigator, Solrun Sigurdardottir, Principal Investigator, Oslo University Hospital
Other Study IDs: 166639
Record Dates: First submitted 2021-12-22; First posted 2022-06-01 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Bardet-Biedl Syndrome
Keywords: Retinitis Pigmentosa; Obesity; Polydactyly; Bardet-Biedl Syndrome; Cognitive deficits
MeSH Terms: conditions — Bardet-Biedl Syndrome; Retinitis Pigmentosa; Obesity; Polydactyly; Cognition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood tests will include renal-, liver-, bone-, lipid-, and endocrine profiles. EDTA blood samples will be sent to Telemark hospital for genetic testing, for individuals lacking molecular genetic confirmation of diagnosis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Bardet-Biedl syndrome (BBS; OMIN #209900) is a rare genetic disorder characterized by six core features: rod-cone dystrophy (retinitis pigmentosa), polydactyly, obesity, genital anomalies, renal anomalies, and learning difficulties. This study aims to contribute to genetic and medical knowledge of BBS, and to provide information on quality of life in adults with BBS and their close relatives. Participants will undergo medical assessments (ocular, oral, and physical examinations) and self-reporting of quality of life, diet, cognitive and emotional symptoms. There are some known genotype-phenotype associations in BBS and participants will be offered genetic testing. It is important to map both genotype and associated phenotype in order to provide optimal treatment and follow-up. Individuals with BBS, age 16 years or older, will be invited to participate. The investigators expect to enroll at least 25 male and female adults with BBS and 15 of their parents to participate in qualitative interviews. These interviews will investigate parents' experiences having a child with BBS, satisfaction with health care services, experience with social and family life, and psychological health.

DETAILED DESCRIPTION:
Improved care for adults with BBS living in Norway necessitates increased knowledge of pertinent health-related, emotional, and educational, employment and psychosocial issues. Adults with BBS living in Norway may face new challenges and have unmet healthcare needs. Therefore, the investigators intend to evaluate the adult with BBS as a person with special needs (e.g. need for support systems, lack of social opportunities, and mental health problems) and long-term challenges.This project will describe the visual, medical, physical, nutritional, and psychological difficulties experienced by people with BBS. The planned multi-disciplinary clinical evaluation in this study can help address the existing knowledge gaps. Relatives who help their loved ones with various activities of daily living may experience reduced quality of life and altered social roles. Therefore, the investigators also want to study the quality of life and psychological status of close relatives. This project might contribute information for new clinical protocols and suggest areas for further research in genetics, healthcare needs and quality of life for people living with BBS.

ELIGIBILITY:
Inclusion Criteria:

Individuals diagnosed with BBS (see below), age 16 years or older. BBS is characterized by six core features : rod-cone dystrophy (retinitis pigmentosa), polydactyly, obesity, genital anomalies, renal anomalies, and learning difficulties.

Additional features include speech delay, developmental delay, diabetes mellitus, dental anomalies, congenital heart disease, brachydactyly (shortening of fingers/toes), ataxia, and anosmia/hyposmia (deficienct sense of smell). A minimum of four of the core features, or three core features and two additional features are required for the clinical diagnosis of BBS.

Exclusion Criteria:

Individuals age < 16 years, current severe illness or known diagnosis of autism.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with BBS, age 16 years or older
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
The Medical Outcome Study 36-item Short Form Health Survey (SF-36) | Feb 2022-Dec 2026
  Health related quality of life (HRQOL) including measures of Physical and mental HRQOL. The SF-36 is a generic quality of life scale which has been validated in Norway. SF-36 evaluates eight domains of health: physical functioning, role limitation due to physical problems, bodily pain, general perception of health, social functioning, role limitations due to emotional functioning, vitality and mental health. Items on each scale are summed to yield a score from 0-100. A higher score means better quality of life. A license from Quality Metric is used for scoring (License number QM051240). The eight domains are summarized into physical component summary scores and mental component summary scores.
Needs and Provision Complexity Scale | Feb 2022-Dec 2026
  Presence of health care needs. This is an interview that evaluates the needs for healthcare and social support services. It has two parts: Part A (Needs) is completed by the clinician to evaluate each patient's need for health and social care; and Part B (Gets) is to evaluate to which these needs are met through the services that have been provided, based on information provided by the patient and a close relative. Each part includes 15 items with a total scoring range of 0-50 covering low and high levels of needs. There are six subscales representing two domains: Health and personal care needs, and Social and support needs. This scale was developed in the UK for neurological conditions and has been translated and used in Norway.
Behavioral Rating Inventory of Executive Function- Adult Version | Feb 2022-Dec 2026
  Assessing cognitive problems. BRIEF-A is a measure of everyday executive functions using self-reports. It includes 75 items that assess nine aspects of executive functioning symptoms of everyday life. Raw scores are transformed into age-corrected T-scores. Higher T-scores mean better executive function.

SECONDARY OUTCOMES:
Short Physical Performance Battery; | Feb 2022-Dec 2026
  Assessing physical problems. This is a group of measures that combines the results of the gait speed, chair stand and balance tests. The scores range from 0 (worst performance) to 12 (best performance).It has been used as a predictive tool for possible disability.
The Hospital Anxiety and Depression Scale; | Feb 2022-Dec 2026
  Assessing anxiety and depression symptoms. This is a generic instrument used to address symptoms of depression and anxiety. The two subscales (anxiety, depression) consist of seven items rated on a four-point scale from 0 (no symptom) to three (severe symptom). A score of >7 on either subscale indicates at least a mild level of depressive or anxiety symptoms. A total HADS score may be used as a global measure of psychological distress. It is widely used in various somatic and psychiatric populations.
Three Factor Eating Questionnaire-R21 | Feb 2022-Dec 2026
  Assessing eating habits. This is a frequently used validated scale that measures three domains of eating behavior (cognitive restraint, uncontrolled eating and emotional eating). The first 20 items are rated on a 4-point Likert scale and the item 21 is answered through an 8-point Likert scale. Scores range from 0-100, with higher scores being indicative of greater restraint eating.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte von der Lippe, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Norwegian BBS patients belong to a small group. Access to a limited version of the dataset containing selected variables may be made available on request.

REFERENCES:
- [Derived] Rustad CF, Bragadottir R, Nordgarden H, Miller JU, Weedon-Fekjaer MS, Arfa S, Asten PM, Tveten K, von der Lippe C, Sigurdardottir S. Healthcare needs, care use and health status outcomes in adults with Bardet-Biedl syndrome: a cross-sectional study in Norway. BMJ Open. 2025 Apr 22;15(4):e095986. doi: 10.1136/bmjopen-2024-095986. PMID 40262952